CLINICAL TRIAL: NCT03070067
Title: Spectrometry for TIA Rapid Assessment (SpecTRA) Project: Study 2-Validation of Clinical Features and Protein Biomarkers
Brief Title: SpecTRA; A Study of the Validation of Protein Biomarkers in Transient Ischemic Attack
Status: Completed | Type: Observational
Sponsor: Andrew Penn (Other)
Collaborators: Genome Canada (Other); Genome British Columbia (Industry); Genome Alberta (Other); Vancouver Island Health Authority (Other); LifeLabs (Unknown); Heart and Stroke Foundation of Canada (Other); Stroke Services BC (Unknown); Bruker Daltonics (Industry); British Columbia Centre for Disease Control (Other Government)
Responsible Party: Sponsor-Investigator, Andrew Penn, Principal Investigator, Vancouver Island Health Authority
Organization: Vancouver Island Health Authority (Other)
Other Study IDs: Island Health CREB C2015-042
Record Dates: First submitted 2017-02-28; First posted 2017-03-03 (Actual); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: TIA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Human plasma collected within 24 hours of symptom onset; MRI; Holter +\- Extended Cardiac Monitoring
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Mild ACVS-definite: Clinical diagnosis of ACVS, and imaging positive (either DWI+ or CT/CTA+).
  Interventions: Other: Non-Interventional Study
- Mild ACVS-possible: Clinical diagnosis of ACVS, and DWI- and/or CTA-.
  Interventions: Other: Non-Interventional Study
- Mimic: Clinical diagnosis of mimic and imaging negative.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — This is a non-interventional study. However, several blood samples will be taken which would not be taken as part of standard of care.

SUMMARY:
A clinical decision support rule/tool for classification of TIA/mimic that will enable rapid detection of ACVS in hyper-acute settings is being developed. Also under development is a multi-protein test using mass spectrometry (MS). This test will provide TIA results within an hour or two for a fraction of the price of neuroimaging. With guidance provided by this test at their disposal, physicians can inform patients whether they can go home safely or whether they need further testing. The right patients will receive the right treatment, reduce unwarranted imaging risks and costs, and reduce the burden of stroke. The Heart and Stroke Foundation will work to ensure that physicians, allied healthcare providers, the public and other stakeholders are aware of the outcomes and clinical impacts of this project.

Further, work is being done to establish the mechanisms to develop a strong phenotype for TIA that includes medical imaging (MRI), cardiac monitoring, cognitive assessments, and surveillance of health outcomes for extended periods of time.

DETAILED DESCRIPTION:
Patients who fulfill all inclusion and none of the exclusion criteria after giving informed consent will be enrolled in the Validation study.

At enrollment, patients will receive a stroke nurse assessment in the Emergency Department (ED) and clinical information documented on an ACVS Assessment Form/SpecTRA Case Report Form. Patients will provide 6 mL of blood drawn into a purple-top EDTA tube that will be processed for proteomic analyses. These blood draws may or may not occur with the standard-of-care blood draw in the ED or stroke unit. Clinical orders include medical imaging (MRI +/- CT/CTA), cardiac monitoring (24hr +/- extended event monitoring). Patients will be referred by the attending ED physician to a stroke clinic for neurological consultation within 48 hours - 7 days, whereby diagnosis of (i) possible ACVS; (ii) definite ACVS or (iii) mimic will be made. At the stroke clinic a cognitive screening test will be administered either as part of usual clinical care by treating physicians, nurses, or a study coordinator. A re- assessment will be repeated at 90 days by phone. MRI will be reviewed initially for clinical interpretation at the neurological consultation for evidence of brain ischemia (DWI+) and later by neuro-radiologists for definitive diagnosis in study purposes. Final adjudication of TIA and aetiology will be done by the non-blinded principal investigators at each site based on diagnostic results plus 90-day and up to 2-year outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Time from the neurologic event to study enrollment is within <24 hours of first symptom onset.
2. All planned diagnostic tests for stroke evaluation must be completed, including brain imaging (MRI) within 4-7 days; and 24-hour +/- extended cardiac monitoring.
3. Be able to provide blood samples collected either under standard-of-care presentation in the ED or hospital-based stroke unit, or by a study-specific personnel outside of standard-of-care collections.
4. Age ≥18 years.
5. Written informed consent consistent with local regulations governing research in human subjects.

Exclusion Criteria:

1. Stroke severity exceeding 4 on the National Institutes of Health Stroke Severity scale (NIHSS <4).
2. Contraindications to brain imaging.
3. Non-English speaking, unless translator present.
4. Isolated monocular blindness.

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population includes individuals presenting to the hospital ED or stroke clinic with symptoms suggesting mild ACVS who would be referred to the outpatient stroke clinic. Patients will be recruited primarily from emergency department settings or hospital-based stroke units.
Sampling Method: Non-Probability Sample
Enrollment: 1150 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Validation of a Protein Classifier for the Diagnosis of TIA in the Emergency Department | 24 Hours
  Calculated score for distinguishing ACVS from Mimic based on previously locked-down formula involving 16 proteins measured using multiple reaction monitoring in blood samples taken within 24 hours from onset of symptoms.

SECONDARY OUTCOMES:
The Validation of a Clinical Classifier for the Diagnosis of TIA in the Emergency Department. | 24 hours
  Calculated score for distinguishing ACVS from Mimic based on previously locked-down formula involving 50 clinical variables recorded on a standardized case report form.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Penn, M.D., Principal Investigator — Vancouver Island Health Authority; Shelagh Coutts, M.D., Principal Investigator — Alberta Health services; Christoph Borchers, P.hD, Principal Investigator — UVic-Genome BC Proteomics Centre
Locations (2):
- Canada (2):
  - Foothills Medical Centre, Calgary, Alberta
  - Vancouver Island Health Authority, Victoria, British Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Penn AM, Croteau NS, Votova K, Sedgwick C, Balshaw RF, Coutts SB, Penn M, Blackwood K, Bibok MB, Saly V, Hegedus J, Yu AYX, Zerna C, Klourfeld E, Lesperance ML. Systolic blood pressure as a predictor of transient ischemic attack/minor stroke in emergency department patients under age 80: a prospective cohort study. BMC Neurol. 2019 Oct 25;19(1):251. doi: 10.1186/s12883-019-1466-4. PMID 31653207